CLINICAL TRIAL: NCT02026973
Title: Impact of Endogenous Estrogen on Somatostatin Inhibition and Growth Hormone Rebound in Older Women
Brief Title: Impact of Endogenous E2 on SSI and GH Rebound
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johannes D. Veldhuis, Professor, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13-007623
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Normal Healthy Volunteers
MeSH Terms: interventions — Fulvestrant; Anastrozole; Somatostatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- IM Placebo/Oral Placebo (Experimental): IM placebo given once on Day 1; Oral placebo pills daily x14-18 days. Somatostatin 1mcg/kg/hr will be administered for 2 hours from 8-10AM on the overnight visit.
  Interventions: Drug: Placebo; Drug: Somatostatin
- IM Placebo/PO Anastrozole (Experimental): IM placebo given once on Day 1; Oral Anastrozole 2.0mg pills daily x14-18 days. Somatostatin 1mcg/kg/hr will be administered for 2 hours from 8-10AM on the overnight visit.
  Interventions: Drug: Anastrozole; Drug: Placebo; Drug: Somatostatin
- IM Fulvestrant/PO Placebo (Experimental): IM Fulvestrant 250mg given once on Day 1; Oral Placebo pills daily x14-18 days. Somatostatin 1mcg/kg/hr will be administered for 2 hours from 8-10AM on the overnight visit.
  Interventions: Drug: Fulvestrant; Drug: Placebo; Drug: Somatostatin
- IM Fulvestrant/IM Anastrozole (Experimental): IM Fulvestrant 250mg given once on Day 1; Oral Anastrozole pills daily x14-18 days. Somatostatin 1mcg/kg/hr will be administered for 2 hours from 8-10AM on the overnight visit.
  Interventions: Drug: Fulvestrant; Drug: Anastrozole; Drug: Somatostatin

INTERVENTIONS:
Drug: Fulvestrant
  Arms: IM Fulvestrant/IM Anastrozole; IM Fulvestrant/PO Placebo
Drug: Anastrozole
  Arms: IM Fulvestrant/IM Anastrozole; IM Placebo/PO Anastrozole
Drug: Placebo
  Arms: IM Fulvestrant/PO Placebo; IM Placebo/Oral Placebo; IM Placebo/PO Anastrozole
Drug: Somatostatin

SUMMARY:
Endogenous estrogens maintain growth hormone (GH) secretion in postmenopausal women by potentiating endogenous GH-releasing hormone (GHRH) drive and restraining somatostatin inhibition of GH release.

DETAILED DESCRIPTION:
Systemic concentrations of testosterone (Te), estradiol (E2), GH, IGF-I and IGFBP-3 decline in healthy aging individuals (1-3). Sex-steroid deprivation accentuates GH and IGF-I depletion, since Te and E2 stimulate GH and IGF-I production in older adults, hypogonadal patients of all ages, and patients undergoing gender reassignment (1,2,4). Tamoxifen blocks the effect of Te, suggesting involvement of E2 in GH's stimulation in men (5). E2 also stimulates GH secretion in women, putatively via the nuclear estrogen receptor (ER-alpha) (1,2,6,7). Because Te, E2 and GH fall with menopause, and Te is converted to E2 by aromatization in the body (8-10), we postulate that diminished Te concentrations, Te→E2 concentrations and low E2 mediate low GH output in older women. What remains unknown is whether the low E2 levels in postmenopausal women retain GH-stimulating effects. To test this notion would require blocking: (i) aromatase-enzyme activity, which mediates E2 synthesis from Te, and/or (ii) estrogen receptor-alpha, which transduces most of E2's stimulation of the GH axis.

ELIGIBILITY:
Inclusion:

1. 60 healthy post-menopausal women (ages 55 to 80 y);
2. BMI 18-30 kg/m2
3. Community dwelling; and voluntarily consenting

Exclusion:

1. Recent use of psychotropic or neuroactive drugs (within five biological half-lives);
2. Obesity (outside weight range above);
3. Laboratory test results not deemed physician acceptable, cholesterol >250, triglycerides > 300, BUN >30 or creatinine > 1.5 mg/dL, liver function tests exceeding twice upper limit of normal, electrolyte abnormality, anemia;
4. Drug or alcohol abuse, psychosis, depression, mania or severe anxiety;
5. Systemic inflammatory disease;
6. Endocrinopathy, other than primary thyroidal failure receiving replacement;
7. Nightshift work or recent transmeridian travel (exceeding 3 time zones within 7 days of CRU admission);
8. Acute weight change (loss or gain of > 2 kg in 6 weeks);
9. Systemic illness
10. Unwillingness to provide written informed consent.
11. Allergy to anastrozole or fulvestrant (treatment drugs).
12. History or suspicion of breast cancer.
13. History of carcinoma (excluding localized basal cell carcinoma removed or surgically treated with no recurrence).
14. History of thrombotic arterial disease (stroke, TIA, MI, angina) or deep-vein thrombophlebitis.
15. History of CHF, cardiac arrhythmias, congenital QT prolongation, and medications used to treat cardiac arrhythmias.
16. Pre-menopausal status as determined by screening hormone measurements.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The summed mass of GH over 10 hours. | 14-18 days: From date of randomization to overnight visit
  Subjects will be given placebo/fulvestrant and placebo/anastrozole on Day 1 to take for 14-18 days. For one night between Days 14-18, from date of randomization, subjects will undergo a 15-h overnight (2200-1300h) fasting, 10-min blood sampling. The primary analytical outcome is the summed mass of GH secreted in pulses over the first 10h of overnight blood samples. Pulsatile GH is relevant, since sex-steroid hormones and regulatory peptides uniquely control GH secretory-burst mass.

SECONDARY OUTCOMES:
The summed mass of GH over a 2h Somatostatin infusion and 3h rebound window | 14-18 days: From date of randomization to overnight visit
  Subjects will be given placebo/fulvestrant and placebo/anastrozole on Day 1 to take for 14-18 days. For one night between Days 14-18, from date of randomization, subjects will undergo a 15-h overnight (2200-1300h) fasting, 10-min blood sampling. The secondary outcome is summed GH secretory-burst-mass values during the overnight visit, specifically: a 2-h somatostatin infusion and subsequent 3-h rebound window.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Veldhuis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States